CLINICAL TRIAL: NCT01297829
Title: Does Preoperative Caldolor Decrease the Requirement for Postoperative Narcotics in Patients Undergoing Laparoscopic or Open Inguinal and/or Umbilical Hernia Repair? A Randomized, Double-Blind, Prospective Trial
Brief Title: Does Preoperative Caldolor Decrease the Requirement for Postoperative Narcotics
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Barnabas Medical Center (Other)
Collaborators: Cumberland Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Ronald S. Chamberlain, Chairman and Chief Department of Surgery, St. Barnabas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2010-11-15
Record Dates: First submitted 2010-11-15; First posted 2011-02-17 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Postoperative Pain
Keywords: ibuprofen; postoperative narcotics; visual analog pain scale; inguinal hernia repair; umbilical hernia repair
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Caldolor (Active Comparator)
  Interventions: Drug: Intravenous Ibuprofen
- Placebo (Placebo Comparator)
  Interventions: Other: IV Placebo

INTERVENTIONS:
Drug: Intravenous Ibuprofen — 800 mg IV ibuprofen 30 minutes preoperatively
  Other Names: Caldolor
  Arms: IV Caldolor
Other: IV Placebo — IV normal saline
  Arms: Placebo

SUMMARY:
Caldolor® is an intravenous (IV) formulation of ibuprofen encompassing analgesic, anti-inflammatory and antipyretic (anti-fever) properties. Caldolor® is the first IV antipyretic approved by the US Food and Drug Administration (FDA), providing an alternate route for administration of ibuprofen when the oral route is not preferable. Recent studies have reported that Caldolor® decreases morphine use and pain at rest and with movement compared to patients not receiving this drug.

The hypothesis of the proposed study is that a single dose of Caldolor® 800 mg given 30 minutes preoperatively for patients undergoing laparoscopic or open inguinal and/or umbilical hernia repair will result in a >20% decrease in postoperative narcotic use within the first 24 hours and at 7 days, and decreased VAS Pain Score at 2 hours, 1 day, 3 days and 7 days after surgery. The use of less postoperative narcotics has been associated with a faster return of normal bowel function and resumption of normal ambulatory status thus resulting in improved general well being for the patient.

ELIGIBILITY:
Inclusion Criteria:

* primary inguinal and/or umbilical hernia repair
* age > 18 years old

Exclusion Criteria:

* history of gastrointestinal bleeding
* allergy to ibuprofen
* creatinine > 1.5 mg/dL

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-02; Primary Completion 2013-08 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative Narcotic Use | 7 days
  Post-operatively, the patient will receive a journal to record daily medication used up to and including post-operative day 7.

SECONDARY OUTCOMES:
Postoperative Visual Analog Pain Scale | 7 days
  The patient will receive a Visual Analog Pain Scale to complete 2 hrs post-operatively, post-operative day 1, post-operative day 3 and post-operative day 7

CONTACTS AND LOCATIONS:
Overall Officials: Ronald S Chamberlain, MD, MPA, FACS, Principal Investigator — St. Barnabas Medical Center
Locations (1):
- Saint Barnabas Medical Center, Livingston, New Jersey, United States